CLINICAL TRIAL: NCT06874231
Title: Clinical Application of a Brain Connectivity Marker for Early Detection of Alzheimer's Disease
Brief Title: Brain Connectivity Marker for Alzheimer's Disease
Acronym: BRAINCONN
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Joana Braga Pereira, Principal Investigator, Karolinska Institutet
Other Study IDs: Dnr 2023-00026-02
Record Dates: First submitted 2023-04-04; First posted 2025-03-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
Keywords: MRI; Cognition; MEG/EEG; Biomarkers
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuroimaging; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid and blood plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- SCI normal: Subjects with subjective cognitive impairment with normal amyloid levels.
  Interventions: Other: Neuroimaging
- SCI abnormal: Subjects with subjective cognitive impairment with low amyloid levels.
  Interventions: Other: Neuroimaging
- MCI abnormal: Subjects with mild cognitive impairment with low amyloid levels.
  Interventions: Other: Neuroimaging
- AD abnormal: Subjects with Alzheimer's disease with low amyloid levels.
  Interventions: Other: Neuroimaging

INTERVENTIONS:
Other: Neuroimaging — The investigators will collect imaging sequence, cognitive test scores, clinical data and biofluid samples
  Other Names: Cognitive assessment

SUMMARY:
The main purpose of this project is to establish whether changes in brain connectivity can be used to predict the development of Alzheimer's disease (AD).

DETAILED DESCRIPTION:
To achieve this aim, the investigators will perform six different studies that have been designed to achieve the following specific objectives:

1.1. Identify changes of brain connectivity in individuals who show abnormal AD amyloid biomarkers in the cerebrospinal fluid and blood.

1.2. To assess the correlation between brain connectivity changes and biomarkers of synaptic dysfunction and inflammation as well as alterations of electrical brain signals.

1.3. Establish whether alterations of brain connectivity could be improved after patients start treatment with cholinesterase inhibitors.

1.4. Assess differences in brain connectivity between patients receiving treatment with statins and those not taking this medication.

1.5. Determine whether brain connectivity changes can predict longitudinal cognitive decline and conversion to AD dementia.

1.6. Assess whether different microorganisms can grow more rapidly in the cerebrospinal fluid from AD patients compared to controls and whether their levels are associated with brain connectivity.

1.7. Evaluate the relationship between brain connectivity and the integrity of the locus coeruleus, which is the earliest site of AD pathology

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for subjects with subjective cognitive complaints:

   * MMSE (Mini-mental test) or MoCA (Montreal Cognitive Assessment) points between 26 and 30.
   * Absence of cognitive impairment.
   * Memory problems reported by the participant/family member.
   * Do not fulfill criteria for mild cognitive impairment or dementia.
   * Must speak and understand Swedish.
2. Inclusion criteria for patients with mild cognitive impairment:

   * MMSE (Mini-mental test) or MoCA (Montreal Cognitive Assessment) points between 24 and 30.
   * Impaired memory function.
   * Do not fulfill criteria for dementia.
   * Must speak and understand Swedish.
   * Must have abnormal cerebrospinal fluid amyloid-β 42/40 ratio levels, which is a biomarker of Alzheimer's disease.
3. Specific inclusion criteria for patients with Alzheimer's disease:

   * MMSE (Mini-mental test) or MoCA (Montreal Cognitive Assessment) points between 18 and 28.
   * Impaired memory function in addition to impaired executive abilities, language function, visuospatial ability and/or attention/psychomotor speed.
   * Meet NINCDS-ADRDA and DSM-IV criteria for probable Alzheimer's disease.
   * Must speak and understand Swedish.
   * Must have abnormal spinal fluid amyloid-β 42/40 ratio levels, which is a biomarker of Alzheimer's disease.

Exclusion Criteria:

* Alcohol or drug abuse.
* Unstable somatic disease or organ failure.
* Refuse to cerebrospinal fluid testing and/or blood sampling, neuropsychological testing, brain imaging, electroencephalogram or magnetoencephalogram.

In addition, participants who have claustrophobia or some form of metal implant in their body that may interfere with the brain imaging scan will be excluded from the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects across the AD continuum
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Brain connectivity can predict the development of Alzheimer's disease | 4 years
  The investigators will build a multilayer network for each patient using DWI and fMRI images, following a methodology similar to that described in Multiplex Connectome Changes Across the Alzheimer's Disease Spectrum Using Gray Matter and Amyloid Data. Specifically, each patient's brain connectivity will be modeled as a multiplex network, where distinct imaging modalities define different layers. The structural connectivity layer will be derived from diffusion-weighted imaging (DWI), capturing white matter fiber tract connections between brain regions. The functional connectivity layer will be built using functional MRI (fMRI), measuring temporal correlations of neural activity across regions. Nodes in the network will correspond to anatomically defined brain regions, and inter-layer edges will be established to link homologous regions across layers, enabling integration of structural and functional information.

SECONDARY OUTCOMES:
Relationship between multilayer connectivity and other imaging sequences, cognition and biofluid biomarkers | 4 years
  The investigators will measure the association between multilayer brain connectivity with biomarkers and clinical measures from the participants, including markers of amyloid, tau, vascular pathology and tests measuring memory, executive function, language and visuospatial skills. These analyses will be conducted using linear regression and linear mixed effects models for longitudinal outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No